CLINICAL TRIAL: NCT00893464
Title: An Open-Label, Dose-Escalation, Phase 1 Study of IXAZOMIB (MLN9708), A Second-Generation Proteasome Inhibitor, in Adult Patients With Lymphoma
Brief Title: A Study of IXAZOMIB in Adult Patients With Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C16002; U1111-1166-8981 (Registry Identifier: WHO (UTN))
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IXAZOMIB (Experimental)
  Interventions: Drug: IXAZOMIB

INTERVENTIONS:
Drug: IXAZOMIB — Patients will be administered IXAZOMIB by IV on Days 1, 8, and 15 of a 28-day cycle. The first stage of the study will be initiated at a starting dose of 0.125 mg/m2. Subsequent doses will increase until a maximum tolerated dose (MTD) is established.

SUMMARY:
This study is an open-label, multicenter, phase 1, dose-escalation study of IXAZOMIB in adult patients with lymphoma. This study will be the first to administer IXAZOMIB to patients with lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years or older.
2. Eastern Cooperative Oncology Group performance status 0-2.
3. Patients must have a confirmed diagnosis of lymphoma that is relapsed and/or refractory after at least 2 prior chemotherapeutic regimens and for which no curative option exists. Patients with Waldenstrom's macroglobulinemia are not eligible for enrollment in this study. Patients with Hodgkin lymphoma are considered eligible for this study.
4. Suitable venous access for PK and pharmacodynamic evaluations.
5. Female patients who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse.

   Male patients who agree to to practice 2 effective methods of contraception or abstain from heterosexual intercourse.
6. Voluntary written consent must be obtained.
7. Adequate blood and chemistry values during the screening period:

   * Absolute neutrophil count (ANC) ≥ 1,500/mm3; platelet count ≥ 100,000/mm3.
   * Total bilirubin must be ≤ 1.5 × the upper limit of the normal range upper limit of normal (ULN).
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) must be ≤ 2.5 × the upper limit of normal (ULN). AST and ALT may be elevated up to 5 times the upper limit of normal if their elevation can be reasonably ascribed to the presence of metastatic disease.
   * Calculated creatinine clearance ≥ 30 mL/minute.

Exclusion Criteria:

1. Peripheral neuropathy ≥ Grade 2.
2. Female patients who are lactating or have a positive serum pregnancy test during the screening period .
3. Major surgery within 14 days before the first dose of treatment.
4. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before the first dose of study treatment.
5. Life-threatening illness unrelated to cancer.
6. Diarrhea > Grade 1 based on the NCI CTCAE categorization.
7. Systemic antineoplastic therapy/or radiotherapy within 21 days before the first dose of study treatment.
8. Systemic treatment with prohibited medications.
9. Patient has symptomatic brain metastases.
10. Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or myocardial infarction within the past 6 months.
11. QTc > 470 milliseconds (msec) on a 12-lead electrocardiogram (ECG) obtained during the screening period.
12. Known human immunodeficiency virus (HIV), hepatitis B or hepatitis C positive.
13. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
14. Treatment with any investigational products within 28 days before the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (7):
- United States (6):
  - Tower Cancer Research Center, Beverly Hills, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Kansas University Medical Center, Westwood, Kansas
  - Cornell University, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Wisconsin Madison, Madison, Wisconsin
- Jewish General Hospital, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in the United States and Canada from 20 August 2009 to 23 October 2014. Out of a total of 31 participants who were enrolled, 30 participants received at least 1 dose of ixazomib.
Pre-assignment Details: Participants with historical diagnosis of lymphoma, for whom at least 2 previous chemotherapeutic regimens failed and no curative option existed enrolled in 1 of 8 treatment groups based on ixazomib's dose: 0.125 milligram per square meter (mg/m^2), 0.25 mg/m^2, 0.5 mg/m^2, 1 mg/m^2, 1.4 mg/m^2, 1.76 mg/m^2, 2.34 mg/m^2, 3.11 mg/m^2.
Groups:
- Ixazomib 0.125 mg/m^2: Ixazomib (MLN9708) 0.125 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until progressive disease (PD) or unacceptable toxicity.
- Ixazomib 0.25 mg/m^2: Ixazomib (MLN9708) 0.25 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
- Ixazomib 0.5 mg/m^2: Ixazomib (MLN9708) 0.5 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
- Ixazomib 1.0 mg/m^2: Ixazomib (MLN9708) 1.0 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
- Ixazomib 1.4 mg/m^2: Ixazomib (MLN9708) 1.4 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
- Ixazomib 1.76 mg/m^2: Ixazomib (MLN9708) 1.76 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
- Ixazomib 2.34 mg/m^2: Ixazomib (MLN9708) 2.34 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
- Ixazomib 3.11 mg/m^2: Ixazomib (MLN9708) 3.11 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
Period: Overall Study
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib 1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Started | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5
Completed | 1 | 1 | 1 | 1 | 4 | 7 | 8 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Did not complete therapy/experience PD | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Groups:
- Ixazomib 0.125 mg/m^2: Ixazomib (MLN9708) 0.125 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
- Ixazomib 1.4 mg/m^2: Ixazomib (MLN9708)1.4 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib 1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 | 43.0 | 65.0 | 53.0 | 69.8 (6.18) | 44.7 (16.52) | 64.2 (9.51) | 53.2 (18.51) | 57.1 (15.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1 | 3 | 5 | 1 | 11
  Male | 1 | 1 | 1 | 0 | 3 | 4 | 5 | 4 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White | 0 | 1 | 0 | 1 | 4 | 5 | 9 | 4 | 24
  Black or African American | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5 | 30
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 0 | 0 | 0 | 0 | 5 | 5 | 2 | 12
  United States | 1 | 1 | 1 | 1 | 4 | 2 | 5 | 3 | 18
Body surface area (BSA) [Mean (Standard Deviation); unit: square meter] | 1.890 | 1.840 | 2.430 | 2.000 | 2.100 (0.3445) | 1.811 (0.2183) | 1.830 (0.2403) | 1.960 (0.1785) | 1.911 (0.2534)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 157.0 | 180.0 | 175.0 | 173.0 | 172.8 (13.67) | 168.1 (9.48) | 164.5 (12.87) | 174.2 (9.63) | 169.0 (11.26)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 82.00 | 67.80 | 121.00 | 83.30 | 92.60 (24.148) | 70.70 (13.860) | 73.85 (15.321) | 79.84 (11.436) | 78.57 (17.558)
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG performance status is used to assess how the disease affects the daily living abilities of the participant. It ranges on the scale from 0-5 (0= normal activity; 1= symptoms but ambulatory; 2= in bed for less than (<) 50 percent (%) of the time; 3= in bed for greater than (>) 50% of the time; 4= 100% bedridden; 5= dead.
  participants
    0 | 1 | 0 | 0 | 1 | 2 | 5 | 1 | 3 | 13
    1 | 0 | 1 | 1 | 0 | 2 | 2 | 9 | 2 | 17
Ann Arbor Stage [Number; unit: participants] — Ann Arbor staging is staging system for lymphomas. The stage is determined by location of tumor. Stage I (located in a single region, usually 1 lymph node and surrounding area), Stage II (located in 2 separate regions, an affected lymph node or organ and a second affected area, and both affected areas are confined to 1 side of diaphragm), Stage III (spread to both sides of diaphragm, including organ/area near lymph nodes/spleen), Stage IV (diffuse or disseminated involvement of 1 or more extra lymphatic organs, including any involvement of liver, bone marrow or nodular involvement of lungs).
  participants
    I | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
    II | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 6
    III | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 4
    IV | 0 | 0 | 0 | 1 | 1 | 4 | 4 | 0 | 10
    Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 4
    Not Applicable | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4
Disease Histological Class [Number; unit: participants] — For this outcome measure, number of participants evaluable were 1, 1, 1, 1, 4, 7, 9 and 4 for each arm, respectively.
  participants
    Follicular lymphoma | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 2 | 11
    Diffused large B-cell lymphoma | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 5
    Peripheral T-cell lymphoma not otherwise specified | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 4
    Hodgkin's lymphoma | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
    Others | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
    Cutaneous T-cell lymphoma | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Time Since Primary Diagnosis to First Dose [Mean (Standard Deviation); unit: months] | 53.0 | 50.0 | 75.0 | 82.0 | 105.0 (95.81) | 51.9 (36.95) | 57.2 (63.50) | 113.8 (89.85) | 72.8 (65.22)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; or congenital anomaly; or a medically important event.
Time Frame: Baseline up to 30 days after last dose of study drug
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Groups:
- Ixazomib1.76 mg/m^2: Ixazomib (MLN9708) 1.76 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
- Ixazomib 3.11 mg/m²: Ixazomib (MLN9708) 3.11 mg/m^2, injection, intravenously, once weekly on Days 1, 8, and 15 in 28-day treatment cycles until PD or unacceptable toxicity.
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m²
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5
participants
  Adverse Events | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5
  Serious Adverse Events | 0 | 0 | 0 | 0 | 2 | 1 | 4 | 3

2. Primary Outcome: Number of Participants Reporting at Least 1 TEAE Related to Laboratory Assessments
Description: The number of participants with any markedly abnormal standard safety laboratory values collected throughout study. Hematology, clinical chemistry and urinalysis were performed. TEAEs related to laboratory assessment observed at any time-points were reported under 3 system organ classes: blood and lymphatic system disorders, metabolism and nutrition disorders, and investigations.
Time Frame: Baseline and Days 1, 8, and 15 of each treatment cycle (up to Cycle 45)
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib 1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5
participants
  Blood and lymphatic system disorders | 0 | 0 | 1 | 1 | 2 | 4 | 5 | 3
  Metabolism and nutrition disorders | 0 | 0 | 0 | 1 | 3 | 3 | 5 | 4
  Investigations | 0 | 0 | 0 | 0 | 4 | 2 | 4 | 3

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included body temperature, weight, systolic and diastolic blood pressure and heart rate.
Time Frame: Baseline and Days 1, 8, 15 of each treatment cycle up to 45 treatment cycles
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Number; unit: participants
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest dose of ixazomib that generated dose limiting toxicity (DLT) during Cycle 1 in 0 of 3 or 1 of 6 participants. DLT defined as any of the following considered possibly related to therapy by investigator: Grade 4 neutropenia (absolute neutrophil count [ANC] <500 cell per cubic millimeter [cells/mm^3]) for >7 days; Grade 3 neutropenia with fever or infection; Grade 4 thrombocytopenia for >7 days; platelet count <25,000 cells/mm^3; Grade 3 thrombocytopenia with clinically significant bleeding; platelet count <10,000/mm^3; Grade 2 peripheral neuropathy with pain or Grade 3 peripheral neuropathy; >=Grade 3 nausea/emesis, diarrhea controlled by maximal supportive therapy; Grade 3 QTc prolongation>500 millisecond (msec);any >=Grade 3 nonhematologic toxicity except arthralgia/myalgia; <1 week fatigue; delay in the initiation of the subsequent therapy cycle by >=7 days ; other Grade 2 ixazomib-related nonhematologic toxicities requiring therapy discontinuation.
Time Frame: Treatment Cycle 1
Population: DLT-Evaluable Population included participants who received all Cycle 1 doses of MLN9708 and who completed Cycle 1. If Cycle 1 was interrupted by a DLT, the participant was included in this population.
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants who received ixazomib (MLN9708) 0.125 mg/m^2, 0.25 mg/m^2, 0.5 mg/m^2, 1.0 mg/m^2, 1.4 mg/m^2, 1.76 mg/m^2, 2.34 mg/m^2 or 3.11 mg/m^2 in dose-escalation cohorts .
Arm/Group | All Participants
Number analyzed (Participants) | 28
mg/m^2 | 2.34

5. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: The RP2D of Ixazomib was determined in Part 1 (dose escalation) on the basis of the totality of safety, tolerability, pharmacokinetics (PK), pharmacodynamic and preliminary efficacy data observed in Cycles 1 and 2 and beyond.
Time Frame: Baseline up to Treatment Cycle 45
Population: Safety population included all participants who received at least 1 dose of ixazomib.
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants who received MLN9708 at dose 0.125 mg/m^2, 0.25 mg/m^2, 0.5 mg/m^2, 1.0 mg/m^2, 1.4 mg/m^2, 1.76 mg/m^2, 2.34 mg/m^2 and 3.11 mg/m^2 in Phase 1.
Arm/Group | All Participants
Number analyzed (Participants) | 30
mg/m^2 | 2.34

6. Secondary Outcome: C0: Initial Plasma Concentration After Bolus Intravenous Administration
Description: C0 is the plasma drug concentration at time zero following bolus intravenous injection, obtained from the plasma concentration-time curve.
Time Frame: Cycle 1 Days 1 and 15: Predose and at multiple time points (up to 336 hours postdose)
Population: The pharmacokinetic (PK) analysis population included all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of PK parameters where Days 1 and 15 assessments were available.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5
nanogram per milliliter (ng/mL)
  Day 1 (n= 1, 1, 1, 0, 4, 7, 10, 5) | 7.430 | 59.400 | 106.000 | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 713.883 (149.8808) | 541.771 (292.5175) | 898.461 (370.7638) | 961.205 (410.3423)
  Day 15 (n= 0, 0, 1, 1, 4, 3, 7, 2) | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 56.300 | 383.000 | 497.189 (138.7405) | 499.027 (240.4184) | 802.825 (1658.3231) | 1191.973 (120.2082)

7. Secondary Outcome: AUC(0-168): Area Under the Plasma Concentration-Time Curve From Time 0 to 168 Hours Postdose for Ixazomib
Description: AUC(0-168) is a measure of the area under the plasma concentration time-curve from time 0 to 168 hours postdose
Time Frame: Cycle 1 Days 1 and 15: Predose and at multiple time points (up to 168 hours postdose)
Population: The PK analysis population included all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of PK parameters where Days 1 and 15 assessments were available. AUC(0-168) is not reported for ixazomib 0.125 and 0.25 mg/m^2 as the participants were not evaluable for this parameter.
Measure: Geometric Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 4 | 7 | 10 | 5
hour*nanogram per milliliter (hr*ng/mL)
  Day 1 (n= 0, 0, 0, 0, 4, 6, 7, 5) |  |  | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 636.8 (195.16) | 821.0 (425.74) | 1058.9 (408.84) | 1683.6 (704.59)
  Day 15 (n= 0, 0, 1, 1, 4, 0, 7, 2) |  |  | 175.0 | 732.0 | 1385.4 (343.64) | NA (NA) — Data are not reported as none of the participants were evaluable in the given group at this time point. | 2108.7 (934.02) | 2537.2 (700.04)

8. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for Ixazomib
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Cycle 1 Day 15: Predose and at multiple time points (up to 336 hours postdose)
Population: The PK analysis population included all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of PK parameters.T1/2 is not reported for ixazomib 0.125 and 0.25 mg/m^2 as the participants were not evaluable for this parameter.
Measure: Geometric Mean (Standard Deviation); unit: hr
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 4 | 3 | 7 | 2
hr |  |  | 292.00 | 146.00 | 209.39 (66.466) | 145.57 (55.749) | 107.58 (20.266) | 108.39 (15.627)

9. Secondary Outcome: Rac: Accumulation Ratio for Ixazomib
Description: Rac was estimated as the ratio of AUC (0-168) on Day 15 and AUC (0-168) on Day 1. AUC (0-168) is the area under the plasma concentration-time curve from time 0 to 168 hours postdose.
Time Frame: Cycle 1 Days 1 and 15: Predose and at multiple time points (up to 168 hours postdose)
Population: The PK analysis population included all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of PK parameters. Rac is reported for ixazomib 1.4, 2.34 and 3.11 mg/m^2 groups only as it could not be estimated for the other dosing groups.
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 0 | 6 | 2
ratio |  |  |  |  | 2.174 (0.1436) |  | 2.267 (0.3352) | 2.113 (0.1344)

10. Secondary Outcome: Ae (0-4): Amount of Drug Excreted in Urine From 0 to 4 Hours Postdose
Description: Ae (0-4) is the total amount of drug excreted in the urine from 0 to 4 hours postdose.
Time Frame: Cycle 1, Days 1 and 15: 0 to 4 hours postdose
Population: The PK analysis population included all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of PK parameters where Days 1 and 15 assessments were available.
Measure: Geometric Mean (Standard Deviation); unit: nanogram
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5
nanogram
  Day 1 (n= 1, 1, 1, 0, 4, 6, 8, 5) | 0 | 1440 | 0 | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 8584.4 (5225.23) | 17963.7 (25934.93) | 9897.8 (14935.19) | 25710.4 (22587.05)
  Day 15 (n= 0, 1, 1, 1, 4, 3, 7, 2) | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 661.0 | 568.0 | 10200 | 16711.7 (17064.66) | 17982.2 (18579.76) | 13128.2 (16781.50) | 40712.9 (7424.62)

11. Secondary Outcome: Fe (0-4): Fraction of Dose Excreted Unchanged in Urine From 0 to 4 Hours Postdose
Description: Fe (0-4) is the fraction of the dose excreted unchanged in the urine from 0 to 4 hours postdose, calculated as percentage of the exact dose administered.
Time Frame: Cycle 1, Days 1 and 15: 0 to 4 hours postdose
Population: The PK analysis population was defined as participants who had sufficient dosing data and ixazomib concentration-time data to permit the calculation of PK parameters where Days 1 and 15 assessments were available.
Measure: Geometric Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 7 | 10 | 5
percentage of dose
  Day 1 (n= 1, 1, 1, 0, 4, 6, 8, 5) | 0 | 0.30700 | 0 | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 0.29842 (0.205616) | 0.56896 (0.957931) | 0.23683 (0.433366) | 0.42394 (0.416424)
  Day 15 (n= 0, 1, 1, 1, 4, 3, 7, 2) | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 0.14100 | 0.04900 | 0.53600 | 0.58105 (0.652303) | 0.55331 (0.617730) | 0.31852 (0.481036) | 0.65344 (0.038184)

12. Secondary Outcome: CLr: Renal Clearance
Description: CLr is the volume of plasma from which the drug is completely removed by the kidney in a given amount of time, calculated as the amount of drug excreted in the urine divided by the area under the plasma concentration-time curve, expressed in liter per hour (L/hr).
Time Frame: Cycle 1, Days 1 and 15: 0 to 4 hours postdose
Population: The PK analysis population included all participants who had sufficient dosing data and ixazomib concentration-time data to permit calculation of PK parameters where Days 1 and 15 assessments were available. CLr is not reported for ixazomib 0.125 and 0.25 mg/m^2 as the participants were not evaluable for this parameter.
Measure: Geometric Mean (Standard Deviation); unit: L/hr
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 0 | 0 | 1 | 1 | 4 | 7 | 10 | 5
L/hr
  Day 1 (n= 0, 0,1, 0, 4, 6, 8, 5) |  |  | 0.000000 | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 0.057058 (0.0502156) | 0.118686 (0.177096) | 0.044828 (0.046412) | 0.085303 (0.0539104)
  Day 15 (n= 0, 0, 1, 1, 4, 3, 6, 2) |  |  | 0.024200 | 0.080500 | 0.098174 (0.1041236) | 0.098459 (0.1363057) | 0.034181 (0.0683205) | 0.085569 (0.0121622)

13. Secondary Outcome: Emax: Maximum Observed Effect for Ixazomib
Description: Emax is the maximum inhibition of 20S proteasome activity in whole blood.
Time Frame: Cycle 1 Days 1 and 15: Predose and at multiple time points (up to 168 hours postdose)
Population: The pharmacodynamic analysis population included participants who had sufficient dosing data and effect-time data to permit calculation of pharmacodynamic parameters where Days 1 and 15 assessments were available.
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib 1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 7 | 5 | 4
percentage of inhibition
  Day 1 (n= 1, 1, 1, 1, 3, 7, 5, 4) | 5.150 | 18.500 | 33.200 | 50.500 | 66.333 (14.8352) | 72.186 (8.1009) | 81.860 (3.1801) | 80.200 (3.5618)
  Day 15 (n= 0, 1, 1, 1, 3, 3, 4, 2) | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 64.300 | 19.200 | 44.400 | 69.800 (10.5698) | 74.833 (4.4970) | 79.625 (4.9081) | 83.650 (1.9092)

14. Secondary Outcome: TEmax: Time to Maximum Observed Effect (Emax) for Ixazomib
Description: TEmax: Time to reach the maximum observed effect (Emax), equal to time (hours) to Emax.
Time Frame: Cycle 1 Days 1 and 15: Predose and at multiple time points (up to 168 hours postdose)
Population: as for outcome 13
Measure: Median (Full Range); unit: hr
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib 1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 3 | 7 | 5 | 4
hr
  Day 1 (n= 1, 1, 1, 1, 3, 7, 5, 4) | 0.25000 [0.2500 to 0.2500] | 0.08330 [0.0833 to 0.0833] | 0.10000 [0.1000 to 0.1000] | 0.08330 [0.0833 to 0.0833] | 0.11700 [0.1000 to 0.1330] | 0.08330 [0.0833 to 0.1000] | 0.08330 [0.0833 to 0.2500] | 0.10850 [0.0833 to 0.5330]
  Day 15 (n= 0, 1, 1, 1, 3, 3, 4, 2) | NA — Data are not reported as none of the participants were evaluable in the given group at this time point. | 0.10000 [0.1000 to 0.1000] | 0.10000 [0.1000 to 0.1000] | 0.08330 [0.0833 to 0.0833] | 0.08330 [0.0833 to 0.0833] | 0.08330 [0.0333 to 0.0833] | 0.16665 [0.0833 to 0.2500] | 0.10015 [0.0833 to 0.1170]

15. Secondary Outcome: Overall Best Response
Description: Overall best response is the best response observed for a participant during the study based on International Working Group (IWG) Response Criteria for malignant lymphoma. Complete response (CR) as per IWG is complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. Partial response (PR) is a minimum of 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses and no increase in the size of other nodes. Stable disease (SD) is when a participant fails to attain the criteria needed for a CR or PR, but does not fulfill those for PD. PD is any new lesion or increase by >50% of previously involved sites from nadir.
Time Frame: Baseline up to Cycle 45
Population: Response-evaluable population included participants who received at least 1 dose of study drug, had measurable disease at baseline, and at least 1 postbaseline disease assessment for analyses of response.
Measure: Number; unit: participants
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib 1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4 | 7 | 8 | 3
participants
  CR | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
  SD | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0
  PD | 1 | 1 | 0 | 1 | 2 | 4 | 4 | 2

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug. All AEs/SAEs were reported after administration of the first dose of the study drug and through 30 days after the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Ixazomib 0.125 mg/m^2 | Ixazomib 0.25 mg/m^2 | Ixazomib 0.5 mg/m^2 | Ixazomib 1.0 mg/m^2 | Ixazomib 1.4 mg/m^2 | Ixazomib 1.76 mg/m^2 | Ixazomib 2.34 mg/m^2 | Ixazomib 3.11 mg/m^2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 2/4 | 1/7 | 4/10 | 3/5
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 1/1 | 4/4 | 7/7 | 10/10 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib 0.125 mg/m^2 (N=1) | Ixazomib 0.25 mg/m^2 (N=1) | Ixazomib 0.5 mg/m^2 (N=1) | Ixazomib 1.0 mg/m^2 (N=1) | Ixazomib 1.4 mg/m^2 (N=4) | Ixazomib 1.76 mg/m^2 (N=7) | Ixazomib 2.34 mg/m^2 (N=10) | Ixazomib 3.11 mg/m^2 (N=5)
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 (0) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib 0.125 mg/m^2 (N=1) | Ixazomib 0.25 mg/m^2 (N=1) | Ixazomib 0.5 mg/m^2 (N=1) | Ixazomib 1.0 mg/m^2 (N=1) | Ixazomib 1.4 mg/m^2 (N=4) | Ixazomib 1.76 mg/m^2 (N=7) | Ixazomib 2.34 mg/m^2 (N=10) | Ixazomib 3.11 mg/m^2 (N=5)
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 2 | 6 | 4 | 3
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 5 | 2
Chills (General disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mass (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 3 | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 3
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 4 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 4 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypouricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin fibrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Computerised tomogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photopsia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.